CLINICAL TRIAL: NCT07231094
Title: A Clinical Study Evaluating the Safety, Tolerability, Preliminary Efficacy and Immunogenicity of a Tumor Vaccine Injection Targeting Stressinducible Proteins MICA/B in Combination With the AG Regimen in Patients With Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SapDM275 vaccine Injection
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer Metastatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SapDM275 Tumor Vaccine Injection (Experimental): SapDM275 tumor vaccine was administered via intramuscular injection on Days 1, 15, and 29, once every two weeks.
  Interventions: Biological: SapDM275 Tumor Vaccine Injection

INTERVENTIONS:
Biological: SapDM275 Tumor Vaccine Injection — SapDM275 tumor vaccine was administered via intramuscular injection on Days 1, 15, and 29, once every two weeks.

SUMMARY:
Study design:

This is a single-arm, open-label, dose-escalation and dose-expansion clinical study to evaluate the safety and efficacy of multiple doses of SapDM275 tumor vaccine injection in combination with the AG regimen for the treatment of patients with metastatic pancreatic cancer who have not received prior systemic anti-cancer therapy and are planned to receive AG as first-line treatment.

Treatment must be initiated within 7 days after enrollment. Patients will receive intramuscular injections of SapDM275 tumor vaccine combined with AG regimen until the occurrence of any of the following: disease progression, intolerable toxicity, death (whichever occurs first), the investigator's assessment that the subject is no longer suitable for further treatment, or withdrawal of consent by the subject.

DETAILED DESCRIPTION:
The dose escalation stage inclues two dose cohorts: 5×10⁶active particles and 5×10⁷active particles. Subjects in each cohort will receive a fixed dose via intramuscular injection on Day 1, Day 15, and Day 29.

The traditional3+3 dose-escalation design will be applied:

Three subjects will be enrolled in each cohort. If no dose-limiting toxicity (DLT) is observed during the 35-day observation period, escalation to the next dose level will proceed.

If two or more subjects experience DLTs, dose escalation will be terminated. If one subject experiences a DLT, three additional subjects will be enrolled at the same dose level.

If no DLT occurs in these additional three subjects, escalation to the next dose level will proceed.

If one DLT occurs among the additional three subjects, dose escalation will be terminated.

Dose expansion stage When the high-dose group (5×107 active particles group) in the dose escalation stage achieve good safety profile, a further expansion stage is expected includes a total of approximately 10 subjects (including those in the dose escalation stage).

When ≥2/6 of the patients in the high-dose group (5×107 active particles group) developed DLT during the dose escalation stage, further expansion will return to the low-dose group (5×106 active particles group). The low-dose group could reach a total of approximately 10 subjects (including subjects in the dose escalation stage).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically or cytologically confirmed unresectable metastatic pancreatic cancer;
3. No prior systemic anti-tumor therapy for metastatic pancreatic cancer. Neoadjuvant or adjuvant therapy is permitted, provided no disease progression occurred within 6 months after the last administration;
4. At least one measurable lesion according to RECIST v1.1 criteria;
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
6. Expected survival ≥6 months and ability to receive tumor vaccine and AG regimen treatment;
7. Adequate organ and bone marrow function at screening, defined as follows:

   Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L without granulocyte colony-stimulating factor support; Platelet count (PLT) ≥100 × 10⁹/L without transfusion; Hemoglobin ≥90 g/L; Serum creatinine ≤1.5 × upper limit of normal (ULN) or creatinine clearance ≥50 mL/min (calculated using the Cockcroft-Gault equation); Total bilirubin (BIL) ≤1.5 × ULN; Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≤2.5 × ULN (≤5 × ULN for patients with liver metastases); Coagulation parameters: prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 × ULN; international normalized ratio (INR) ≤1.5 × ULN.
8. Left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiography (ECHO) or multigated acquisition (MUGA) scan;
9. Willingness and ability to provide written informed consent and comply with protocol-specified visits and procedures;
10. Fertile patients (male and female) must agree to use reliable contraception (hormonal, barrier methods, or abstinence) during the study.

Exclusion Criteria:

1. Active or prior autoimmune disease, immunodeficiency, or primary immunodeficiency (including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis). Exceptions include:

   Autoimmune hypothyroidism controlled with thyroid hormone replacement therapy; Well-controlled type 1 diabetes managed with insulin; Eczema, psoriasis, neurodermatitis, or vitiligo limited to skin involvement, with rash <10% of body surface area, stable at baseline, requiring only low-potency topical corticosteroids, and no acute exacerbations within the past 12 months.
2. Receipt of systemic immunosuppressive drugs (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-TNF agents, etc.) within 2 weeks before initiation of study treatment, or anticipated need during the study, except in the following cases:

   Short-term, low-dose systemic immunosuppression or a single pulse dose (e.g., glucocorticoids for 48 hours due to contrast allergy); Use of mineralocorticoids (e.g., fludrocortisone), inhaled corticosteroids, or low-dose corticosteroids (≤10 mg/day prednisone or equivalent) for chronic obstructive pulmonary disease/asthma, or low-dose corticosteroids for orthostatic hypotension/adrenal insufficiency.
3. History of other malignancies within 5 years prior to screening, except for cancers with negligible risk of metastasis or death (5-year recurrence-free survival >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, or stage I endometrial cancer.
4. Severe cardiovascular, cerebrovascular, gastrointestinal, or hepatic disease, including:

   Significant cardiovascular disease within 3 months prior to treatment (e.g., New York Heart Association [NYHA] Class III or IV heart failure, myocardial infarction, or cerebrovascular accident), unstable arrhythmias, or unstable angina; Severe colon or rectal disease, or postoperative complications resulting in grade ≥2 diarrhea, intestinal obstruction, or incomplete obstruction; Clinically significant liver disease, including active viral hepatitis, alcoholic hepatitis or other hepatitis, cirrhosis, hereditary liver disease, or investigator-assessed current alcohol abuse.
5. Active infections requiring treatment, including active HBV or HCV infection; known HIV infection or history of AIDS; active tuberculosis.
6. Toxicities from prior anti-tumor therapies not resolved to grade ≤2 per NCI-CTCAE v5.0 (or higher version) or baseline, except for alopecia and skin hyperpigmentation (any grade allowed).
7. Receipt of a live vaccine within 28 days prior to the first study treatment or planned receipt of a live vaccine during the study.
8. Positive serum pregnancy test or lactating women.
9. History of severe hypersensitivity to biologic products.
10. Any other condition that, in the opinion of the investigator, renders the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
adverse events | From enrollment to the end of treatment at 30 days
  Frequency, number, incidence, and severity of the adverse events and adverse reactions

SECONDARY OUTCOMES:
Objective response rate (ORR) | Every 6 weeks from the first dose of treatment until the date of first documented progression, the start of other treatment, or date of death from any cause, whichever came first, up to 2 years
  Objective response rate will be estimated by CT or MRI depending on the cancer type and location, according to RESIST V1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Hunan, Changsha, China